CLINICAL TRIAL: NCT02949219
Title: A Multicenter Phase II Study of Pembrolizumab (MK-3475) in Patients With Advanced Small Bowel Adenocarcinomas
Brief Title: Pembrolizumab in Treating Patients With Small Bowel Adenocarcinoma That is Metastatic or Locally Advanced and Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU021502I; NCI-2016-01577 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU021502I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Small Intestinal Adenocarcinoma; Recurrent Small Intestinal Carcinoma; Unresectable Small Intestinal Carcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with small bowel adenocarcinoma that has spread to other places in the body or that cannot be removed by surgery. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether pembrolizumab administered to small bowel adenocarcinoma (SBA) patients demonstrates antitumor activity as measured by the confirmed response rate.

SECONDARY OBJECTIVES:

I. To assess survival endpoints (overall survival [OS], progression free survival [PFS]), including stratified analysis by tumor site.

II. To assess whether pembrolizumab is safe in SBA patients by assessing adverse events.

TERTIARY OBJECTIVES:

I. To determine whether PD-L1 expression, as measured by immunohistochemistry (IHC), or microsatellite instability (MSI) status is associated with the response rate overall.

II. To determine if Bim levels in tumor-reactive CD11ahighPD-1+CD8+ peripheral blood T cells can objectively monitor responses to pembrolizumab and to determine if excessive release of soluble B7-H1 (soluble [s]PD-L1) by the tumor leads to Bim upregulation and treatment resistance in SBA.

III. To determine if other tissue-based factors, such as total mutational burden, correlate with response to pembrolizumab.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until disease progression, and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-proven adenocarcinoma of the small bowel at any site (duodenum, jejunum, ileum), excluding ampullary and appendiceal tumors
* Have locally advanced (unresectable) or metastatic small bowel adenocarcinoma
* Willing and able to provide written informed consent for the trial
* Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Had at least one prior line of systemic chemotherapy for metastatic disease; adjuvant therapy would not count toward first-line therapy unless patient recurs less than 6 months after completion of that regimen
* Willing to provide blood and tissue (can be archival) samples for mandatory research purposes
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3 (1.50 x 10^9 /L) obtained =< 28 days prior to registration
* Platelet count >= 100,000/mm^3 (100 x 10^9 /L) obtained =< 28 days prior to registration
* Hemoglobin >= 9.0 g/dL (5.6 mmol/L or 90 g/L) without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) obtained =< 28 days prior to registration
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN obtained =< 28 days prior to registration
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases obtained =< 28 days prior to registration
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance must be >= 60 mL/min for subjects with creatinine levels > 1.5 X ULN using the Cockcroft-Gault formula (glomerular filtration rate [GFR] >= 60 mL/min [1.0 mL/s/m^2] can also be used in place of creatinine or creatinine clearance [CrCl]) obtained =< 28 days prior to registration
* Female subject of childbearing potential have a negative urine or serum pregnancy =< 7 days prior to registration; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * Note: female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Non-adenocarcinoma histology
* Adenocarcinoma originating in the ampulla or appendix; (duodenal tumors that involve the ampulla but originate in the duodenum are eligible)
* Currently participating and receiving study therapy, or have participated in a study of an investigational agent and received study therapy, or used an investigational device =< 4 weeks of registration
* Diagnosis of immunodeficiency or be receiving systemic steroid therapy or any other form of immunosuppressive therapy =< 7 days prior to registration
* History of active TB (bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Any of the following:

  * Prior anti-cancer monoclonal antibody (mAb) =< 4 weeks prior to registration
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy =< 2 weeks prior to registration or who has not recovered to =< grade 1 or baseline from adverse events due to the previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Received major surgery =< 2 weeks prior to registration, subject must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Known additional malignancy that is progressing or requires active treatment or that may interfere with interpretation of response evaluation, in the judgment of the investigator
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging =< 4 weeks prior to registration and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids =< 7 days prior to registration; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Active autoimmune disease (including but not limited to: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn?s disease, patients with a history of symptomatic disease [e.g., rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis (e.g. Wegener?s granulomatosis)]; CNS or motor neuropathy considered of autoimmune origin [e.g., Guillain-Barre syndrome and myasthenia gravis, multiple sclerosis]) that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known history of or any evidence of active, non-infectious pneumonitis
* Active infection requiring systemic therapy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or other immune checkpoint inhibitor (e.g. anti-CTLA4)
* History of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid RNA [qualitative] is detected)
* Received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2024-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McWilliams, Principal Investigator — Academic and Community Cancer Research United
Locations (8):
- United States (8):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab): Patients receive 200 mg pembrolizumab IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 41
Completed | 40
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 30
  More than one race | 0
  Unknown or Not Reported | 3
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 17
    1 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Confirmed Response Rate
Description: The response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients.
Time Frame: 1 year (up to 18 cycles)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 40
percentage of participants | 7.5 [1.6 to 20.4]

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: From study entry to the first of either disease progression or death from any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 40
months | 2.8 [2.7 to 4.2]

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: From study entry to death from any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 40
months | 6.9 [5.1 to 17.1]

4. Secondary Outcome: Number of Participants Who Experienced at Least One Grade 3 or Higher Adverse Events Regardless of Attribution
Description: number of participants who experienced at least one grade 3 or higher adverse events regardless of attribution assessed by National Cancer Institute's Common Terminology Criteria for Adverse Events version 4.03
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 40
Participants | 25

5. Other Pre Specified Outcome: Biomarker Levels
Description: Correlated with clinical data (i.e. response, overall survival, progression free survival, adverse events). These correlations will be done using the Chi-square or Fisher?s exact test for categorical data and Kaplan-Meier methods (including the log-rank test) for the survival endpoints. Univariate Cox regression models will also be done to assess for marker effects on survival endpoints. Descriptive statistics and graphical methods will be used to summarize the data as well. All these analyses will be done overall and by MMR/microsatellite instability status.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 28/40
Serious Adverse Events (participants affected / at risk) | 21/40
Other Adverse Events (participants affected / at risk) | 34/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=40)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Fever (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=40)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (3)
Hyperthyroidism (Endocrine disorders) | 6 (10)
Hypothyroidism (Endocrine disorders) | 11 (45)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (7)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (7)
Localized edema (General disorders) | 1 (9)
Infections and infestations - Oth spec (Infections and infestations) | 1 (2)
Papulopustular rash (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (33)
Alkaline phosphatase increased (Investigations) | 28 (97)
Aspartate aminotransferase increased (Investigations) | 20 (39)
Blood bilirubin increased (Investigations) | 7 (10)
Lymphocyte count decreased (Investigations) | 1 (3)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (6)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT02949219/Prot_SAP_000.pdf